CLINICAL TRIAL: NCT07274293
Title: EVALUATION OF THE TOLERABILITY OF A T-SHIRT CONTAINING PRINTED CERAMICS
Brief Title: EVALUATION OF THE TOLERABILITY AND BIOMEDICAL POTENTIAL OF A GARMENT CONTAINING PRINTED CERAMICS IN MUSCULAR PAIN
Acronym: DZero
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: noiVita Srls (Industry)
Collaborators: University of Eastern Piedmont (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1115/CE; University of Eastern Piedmont (Other: University of Eastern Piedmont)
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Cervical Pain; Lumbar Pain; Muscular; Chronic Pain (Back / Neck); Pain Management
MeSH Terms: conditions — Neck Pain; Low Back Pain; Chronic Pain; Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DZero (Experimental): The DZero product is a new smart fabric containing nanoceramic particles printed on non-compressive elastic fabric, with valuable biomedical and biophysical properties designed to improve human health. It is a non-commercialized, non-invasive medical device that does not release substances onto or into the human body, but achieves its intended use by exploiting body energy. DZero, associated with the manufacturer Noivita s.r.l.s. falls within the category of Class I Medical Devices and is also included in the section ("Miscellaneous Equipment for Physiotherapy and Rehabilitation") in the official database of the Italian Ministry of Health. As a Class I medical device, the manufacturer does not need to involve a notified body for CE marking in the process of demonstrating compliance with the requirements of the MDR, but is itself responsible for issuing the EC declaration of conformity in accordance with Article 19 of the MDR 2017/745, after carrying out the appropriate checks.
  Interventions: Device: DZero

INTERVENTIONS:
Device: DZero — Each person who agreed to participate was given a DZero garment in the form of a T-shirt suitable for their size, so that the garment would fit snugly to the patient's body. The delivery was made by the principal investigator or a specially designated collaborator, who were directly supplied with T-shirts by the Promoter in collaboration with the study manufacturer, who is the direct supplier. The T-shirt was worn for 8 consecutive hours to best express the intrinsic properties related to its components, namely reducing inflammatory conditions and improving muscle tone using body heat. The innovation lies in the engineering of a new smart fabric that, for the first time, integrates nanoceramics and postural structure, exploiting the characteristics of both materials (bioceramics and fabric) to provide significant benefits for improving health and quality of life on a daily basis.

SUMMARY:
Today, a new revolution is underway in the textile industry with the introduction of new technologies that add special functions and properties to fabrics. This innovative revolution will see clothing used not only to protect the body from atmospheric changes or for aesthetic purposes, but also to positively influence health. In this sense, nanoparticles play a key and significant role in this technological evolution as they exhibit exceptional surface properties that allow their effect to be multiplied in comparison to bulky additives and traditional materials. With the development of better technology to deliver pure far infrared radiation (FIR), the benefits of its effects have expanded. The main source of energy needed to power FIR emission from clothing comes from the human body, as it has a higher temperature than the surrounding air. Therefore, energy from the human body is transferred to these ceramic particles, which act as "perfect absorbers," maintaining their temperature at a sufficiently high level and emitting FIR back to the body. At the application level, these fabrics have a wide range of uses, depending on the target of FIR therapy, allowing even in specific conditions to level the concentration of lactic acid, a biological marker associated with cardiovascular diseases and toxins. Other potential benefits include an increase in blood oxygen concentration, improved oxygen and nutrient transport to soft tissues, and muscle relaxation. This potentially prevents contractures while improving muscle tone and alleviating muscle soreness and spasms. This type of tissue approach is a more efficient and less invasive way to provide relief in the area affected by pain, so that it can quickly alleviate muscle pain, cramps, and fatigue, and reduce inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 55;
* Presence of neck or lower back pain for at least 3 months;
* Use of paracetamol in the last 3 months;
* Self-sufficient patients, able to carry out normal daily activities even after wearing the shirt;
* Patients who agree to sign the informed consent form.

Exclusion Criteria:

* Pregnant or breastfeeding patients;
* Presence of chronic malignant diseases;
* Presence of mild/moderate spasticity;
* Use of pharmacological treatments for neuropathic pain (e.g., nicetile, tricyclic antidepressants, opioids, antiepileptics);
* Presence of known severe concomitant brain damage;
* Presence of known concomitant severe brain damage;
* Presence of psychiatric or neurological disorders;
* Presence of tumors or terminal illnesses;
* Alcohol or substance abuse;
* Hypersensitivity to the product;
* Lack of knowledge of the Italian language;
* Participation in other clinical trials in the last 3 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Measuring quality of life | - T0: baseline - T1: after 7 days - T2: after 30 days
  Measuring quality of life, described with the EURO-QoL-5D-5L or EQ-5D-5L. The instrument consists of: a 5-dimensional descriptive system (mobility, self-care ability, habitual activities, pain/discomfort, and anxiety/depression), each of which involves a three-point rating scale (no problem=1 point; some problem=2 points; persistent problem=3 points); and a VAS that requires the subject to answer the question, "How healthy do you feel today?" A score of 0 corresponds to the worst health status ever, while 100 equals the best perceived health level. It is possible to combine the scores of the two sections and determine an overall score.

SECONDARY OUTCOMES:
Measuring the patient's state of well-being | - T0: baseline - T1: after 7 days - T2: after 30 days
  Measurement of well-being described through the Well-Being Index (WHO-5) [23], a self-report tool consisting of 5 statements, to which the subject can respond using a 5-point scale (always=5 points; never=0 points). The total score (from 0 to 25 points) is multiplied by 4 to obtain a score from 0 to 100, where 0 is the worst possible level of well-being and 100 is the best possible level of well-being.
Perceived comfort when wearing DZero | - T0: baseline - T1: after 7 days - T2: after 30 days
  The thermal comfort perceived by the occupants of the environment will also be described, using the ASHRAE (American Society of Heating, Refrigerating and Air-Conditioning Engineers) scale.This scale is a standardized and internationally recognized tool for assessing the subjective thermal comfort of people in a given environment. It is based on a personal assessment expressed on a 7-point scale (from +3, very hot, to -3, very cold, with 0 indicating neither hot nor cold), ranging from a feeling of extreme cold to a feeling of extreme heat.
Measurement of pain perception and its sensory dimensions | -T0: baseline - T1: after 7 days; - T2: after 30 days
  Measurement of pain perception and its sensory dimensions, which were quantified and described using the Short Form-McGill Pain Questionnaire (SF-MPQ). The scale consists of 78 words, each of which describes a painful sensation in detail, divided into four main categories: sensory (sections 1-10), affective (sections 11-15), evaluative (section 16), and miscellaneous (sections 17-20). These 20 sections contain between 3 and 6 descriptive words. The subject to whom it is administered must then highlight the words that best describe their pain. Within each section, the words are assigned a score in ascending order of severity, ranging from 0 (no pain) to 3 (severe), and it is possible to choose more than one word per section; the word corresponding to the highest score will be chosen to define the final score. The words with the highest scores for each section will be added together and used to determine the Pain Rating Index (PRI). The questionnaire only gives a score and not
Assess your perception of fatigue during normal daily activities | -T0: baseline -T1: after 7 days -T2: after 30 days
  Measurement of perceived fatigue and exertion using the Borg scale CR 10. This tool is used to assess the perceived intensity of physical exercise on a numerical scale ranging from 0 (no exertion) to 10 (maximum exertion perceived in one's life). The assessment of perceived exertion is carried out at the end of a daily activity involving at least 30 minutes of movement .This is to avoid the influence of the most recent exertion. It is essential to educate the subject on how to collect data on perceived exertion, avoiding confusion between perceived exertion and perceived pain.

CONTACTS AND LOCATIONS:
Locations (1):
- DAIRI, Alessandria, 15121, Alessandria, Italy

IPD SHARING:
Plan to Share IPD: No